CLINICAL TRIAL: NCT01629173
Title: The Effect of Dynamic Impression Insoles on Plantar Pressure and Pain in Persons With Metatarsal Pain
Brief Title: The Analysis and Applications of Dynamic Impression Insole
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 97-11-12A
Record Dates: First submitted 2011-10-19; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Metatarsalgia
Keywords: plantar pressure; metatarsalgia; insole
MeSH Terms: conditions — Metatarsalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dynamic impression insole (Experimental): We sequentially padded P-cell, Ethylene Vinyl Acetate, and Multiform on the 9-mm thick plastazote under daily walking compression to make dynamic impression insole.
  Interventions: Procedure: Dynamic impression insole
- Custom molded insole (Experimental): The custom molded insole was made by sequentially padded Multiform, P-cell, EVA, and cork on the positive plaster cast impressed by an impression box while holding the subtalar joint at a neutral position.
  Interventions: Procedure: Custom molded insole
- 9-mm uncompressed Plastazote insole (Experimental): We used 9-mm flat Plastazote as an insole
  Interventions: Procedure: 9-mm uncompressed Plastazote
- 7-mm Ethylene Vinyl Acetate (EVA) (Experimental): We used 7-mm flat Ethylene Vinyl Acetate (EVA) as an insole
  Interventions: Procedure: 7-mm Ethylene Vinyl Acetate (EVA)

INTERVENTIONS:
Procedure: Dynamic impression insole — We sequentially padded (1)a 6.5-mm thick P-cell (21 Shore A hardness, Acor orthopedic Inc. Cleveland, Ohio, USA), and (2)a piece of metatarsal pad and arch support made of Ethylene Vinyl Acetate (EVA) (40 Shore A hardness, Schein orthopadie service KG. Remscheid, Germany) to the bottom of the impressed 9-mm thick plastazote (15 Shore A hardness, Schein orthopadie service KG. Remscheid, Germany) with double-sided adhesive tape in the forefoot region and just proximal to the first, second, and third metatarsal head region. We additionally padded a 2-mm thick Multiform (30 Shore A hardness, Schein orthopadie service KG. Remscheid, Germany) on the top of the impressed insole with double-sided adhesive tape.
  Arms: Dynamic impression insole
Procedure: Custom molded insole — The custom molded insole was made by sequentially padded Multiform (30 Shore A hardness, Schein orthopadie service KG. Remscheid, Germany), P-cell (21 Shore A hardness, Acor orthopedic Inc. Cleveland, Ohio, USA), Ethylene Vinyl Acetate (EVA)(40 Shore A hardness, Schein orthopadie service KG. Remscheid, Germany), and cork (50 Shore A hardness, Schein orthopadie service KG. Remscheid, Germany) on the positive plaster cast impressed by an impression box while holding the subtalar joint at a neutral position.
  Arms: Custom molded insole
Procedure: 9-mm uncompressed Plastazote — We used 9-mm flat Plastazote(15 Shore A hardness, Schein orthopadie service KG. Remscheid, Germany) as an insole
  Arms: 9-mm uncompressed Plastazote insole
Procedure: 7-mm Ethylene Vinyl Acetate (EVA) — We used 7-mm flat Ethylene Vinyl Acetate (EVA) (40 Shore A hardness, Schein orthopadie service KG. Remscheid, Germany) as an insole
  Arms: 7-mm Ethylene Vinyl Acetate (EVA)

SUMMARY:
The aim of the study was to investigate the effectiveness of dynamic impression insoles on plantar pressure and pain reduction. A dynamic impression insole was made by sequential padding with Plastazote and P-cell under daily walking compression. The pain levels and plantar pressure with the use of dynamic impression insole were assessed and compared with 7-mm Ethylene Vinyl Acetate (EVA) control, 9-mm uncompressed Plastazote and custom molded insoles. Plantar pressure was measured by a Pedar-X mobile system, and pain level was assessed using a Visual Analog Scales.

DETAILED DESCRIPTION:
Toe deformities may cause prominence of the metatarsal heads (MTH) and distal displacement of fat-pad cushion beneath the MTH, resulting in the metatarsal pain. Foot pain frequently leads to limitation of activities of daily life and deterioration of life quality. Foot orthoses have been commonly used in clinical practice to reduce plantar pressure and subsequent pain. However, the therapeutic efficacies of custom molded insoles with a metatarsal support vary widely with their designs and materials. We designed a simple and effective method that a dynamic impression insole was made by sequential padding of foams with different compressibility under successive dynamic impression in daily walking. A piece of metatarsal pad and arch support made of EVA was attached to the bottom of impressed insole just proximal to the first, second, and third MTH according to the foot impression. Fifty participants with metatarsal pain were recruited from the podiatry outpatient clinic of Taipei Veteran General Hospital. The plantar pressure measurements were carried out under a comfortable and stable walking speed preferred by the participants one month after the dynamic impression and custom molded insoles were well fabricated. All pressure data were processed with the Novel-Win Multimask analysis software. The purposes of this study were to investigate the biomechanics of dynamic impression insole in plantar pressure and pain reduction.

ELIGIBILITY:
Inclusion Criteria:

* Adults with metatarsal pain
* Active in walking without any walking aids

Exclusion Criteria:

* People with flexible flat foot
* Any acute inflammation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in peak plantar pressure value with different insoles | 4 weeks
  We measure peak pressure (in unit of kPa) under forefoot, midfoot, and rearfoot when using different kinds of insoles by Pedar-X mobile in-shoe system (Novel gmbh, Munich, Germany), and data were processed with the Novel-Win Multimask analysis software (Novel gmbh, Munich, Germany) after using dynamic impression insole for four weeks.

SECONDARY OUTCOMES:
Change from baseline in pain levels using Visual Analog Scales | 4 weeks
  We measure pain levels when using different kinds of insoles by Visual Analog Scales after using dynamic impression insole for four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Bao-Chi, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei VGH, Taipei, Taiwan

REFERENCES:
- [Derived] Chang BC, Liu DH, Chang JL, Lee SH, Wang JY. Plantar pressure analysis of accommodative insole in older people with metatarsalgia. Gait Posture. 2014;39(1):449-54. doi: 10.1016/j.gaitpost.2013.08.027. Epub 2013 Aug 31. PMID 24119776